CLINICAL TRIAL: NCT06295744
Title: Patient-Reported Outcomes and Cosmesis Following Five Fraction Whole Breast Irradiation With Simultaneous Integrated Boost
Brief Title: Outcomes and Cosmesis With Whole Breast Irradiation and Boost
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1724; Protocol Version 11/14/2024 (Other: UW Madison); A533300 (Other: UW Madison); UW23114 (Registry Identifier: UWCCC OnCore ID); NCI-2024-01891 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Early-stage Breast Cancer
Keywords: Cosmesis; Simultaneous Integrated Boost; Whole Breast Irradiation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- WBI with SIB (Experimental)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — WBI with SIB delivered over 5 fractions

SUMMARY:
This study is being done to evaluate cosmetic, patient-reported outcome measures (PROMs), and toxicities for women undergoing ultra-short whole breast irradiation (WBI) therapy with simultaneous integrated boost (SIB). 50 participants will be on study for up to 60 months.

DETAILED DESCRIPTION:
The study population will consist of 50 participants with non-metastatic, early-stage invasive breast cancer or ductal carcinoma in situ (DCIS). Eligible patients will include those with a biopsy proven invasive breast cancer or DCIS, greater than or equal to 18 years of age, undergoing breast conserving surgery and adjuvant radiation therapy at UW Health with an indication for WBI with tumor bed boost. Selection need for boost and radiation treatment field design and pre-tx imaging are at the discretion of the treating provider.

Accrual will occur over 5 years at UW Health. Participants will complete 5 treatment visits and 7 study visits over the course of approximately 5.5 years. Research-related outcome measures - MD assessments (e.g., cosmesis) PROMs, and AEs -- will be assessed prior to treatment start, at the 6-week follow-up visit, as well as at 12-, 24-, 36-, 48- and 60-month follow-up visits. Study participation ends after completion of the 60-month follow-up visit.

Objective

• To assess two-year cosmetic outcomes in patients treated with ultra-short WBI with a SIB.

Secondary Objectives

* To assess PROMs via BREAST-Q in patients treated with ultra-short WBI with SIB.
* To assess acute toxicities in patients treated with ultra-short WBI with SIB.
* To assess late toxicities in patients treated with ultra-short WBI with SIB.
* To assess ipsilateral breast tumor recurrence in patients treated with ultra-short WBI with SIB.
* To assess overall survival (OS) in patients treated with ultra-short WBI with SIB.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Histologically confirmed early stage (stage T1-T2) invasive carcinoma of the breast or DCIS
* Breast conserving surgery with negative margins and negative nodes (surgical axillary staging not mandatory), stage N0 or Nx
* Treatment plan should include breast conserving surgery and adjuvant whole breast irradiation (WBI) therapy delivered with 3D-CRT or IMRT techniques
* Treatment plan includes breast tumor bed boost
* Willingness to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Mastectomy of ipsilateral breast
* Lack of histologic diagnosis
* Histologic involvement of the axillary or regional nodes or metastatic disease
* Accelerated partial breast irradiation treatment plan
* Previous history of non-breast malignancy diagnosed in the past 5 years except for basal or squamous cell cancer of the skin
* Previous history of chest radiation therapy
* Previous history of ipsilateral breast cancer
* Concurrent cytotoxic chemotherapy
* Active connective tissue disease including scleroderma
* Inability or unwillingness to return for required follow up visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Harvard Breast Cosmesis Scale Score | up to 2 years post-treatment (treatment ends up to 5 weeks on study)
  4-point scale where 1 is excellent, 2 is good, 3 is fair, and 4 is poor.

SECONDARY OUTCOMES:
Change in BREAST-Q Score | baseline, 6 weeks post-RT, 12 months post-RT, 24 months post-RT, 60 months post-RT (treatment ends up to 5 weeks on study)
  The BREAST-Q questionnaire is scored from 0-100 where higher scores indicate better outcomes in each of 5 domains: Psychosocial Well-Being, Sexual Well-Being, Cancer Worry, Fatigue, and Impact on Work.
Incidence of Acute Toxicities | up to 90 days post-RT (treatment ends up to 5 weeks on study)
  Acute toxicities (including breast dermatitis, induration) will be assessed after final treatment within 90 days of radiation therapy completion using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of Late Toxicities | up to 60 months on study
  Late toxicities (including induration, fibrosis, shrinkage, and telangiectasia) will be assessed greater than 90 days of radiation therapy completion using CTCAE version 5.0
Ipsilateral Breast Tumor Recurrence-Free Survival | up to 60 months on study
  Kaplan-Meier curves will be used to estimate ipsilateral breast tumor recurrence-free survival.
Overall Survival (OS) | up to 60 months on study
  Kaplan-Meier curves will be used to estimate OS.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Schuster, MD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No